CLINICAL TRIAL: NCT01919476
Title: Postprandial Response to Almond Consumption in Overweight Hispanic Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CHO17-ABC
Record Dates: First submitted 2013-07-31; First posted 2013-08-09 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Diabetes, Gestational
Keywords: Postprandial; Insulin resistance; Lipids; Satiety; Almonds
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Meal: Bagel, cream cheese (Active Comparator): Control meal consists of bagel with cream cheese and apple juice.
  Interventions: Other: Bagel; Other: Cream Cheese
- Almond Meal: Bagel, almond butter (Experimental): Almond meal consists of bagel with almond butter and apple juice.
  Interventions: Other: Bagel; Other: Almond Butter

INTERVENTIONS:
Other: Bagel
Other: Cream Cheese
  Arms: Control Meal: Bagel, cream cheese
Other: Almond Butter
  Arms: Almond Meal: Bagel, almond butter

SUMMARY:
Currently, about one third of all women entering pregnancy are obese. The prevalence of metabolic disorders during pregnancy has increased concurrently with the rise in maternal obesity. Although dietary interventions are used routinely to reduce metabolic disease in non-pregnant obese individuals, no specific dietary advice is provided to obese, pregnant women unless they develop gestational diabetes mellitus. In this study, the investigators will specifically assess the effect of replacing dairy fats with almonds in a breakfast meal on the postprandial metabolic response. This cross-over, randomized control trial will examine the postprandial metabolic response to 0 or 2 oz of almonds in standardized test meals in pregnant Hispanic women with prepregnancy BMI between 25 and 40. Hispanics are at higher risk for gestational diabetes and the metabolic syndrome. The investigators hypothesize that consuming almonds in place of dairy fat reduces the glycemic response and improves the postprandial lipid profile in these high-risk women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Hispanic women
* Between 30 and 36 weeks gestation
* Prepregnancy BMI between 25 and 40

Exclusion Criteria:

* Diagnosis of gestational diabetes mellitus
* Preexisting diabetes mellitus
* Renal disease
* Thyroid disease
* Cardiovascular disease
* History of drug abuse
* Nut allergies

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in markers for glucose intolerance. | 0, .5, 1, 2, 3, 4, 5 hours following a meal
  After consuming the breakfast meal markers for glucose intolerance will be measured at the time points listed

SECONDARY OUTCOMES:
Change in metabolic markers | 0, .5, 1, 2, 3, 4, 5 hours following a meal
  After consuming the breakfast meal metabolic markers will be measured at the time points listed.

OTHER OUTCOMES:
Change in satiety markers | 0, .5, 1, 2, 3, 4, 5 hours following a meal
  After consuming the breakfast meal satiety markers will be measured at the time points listed. Satiety questionnaires will also be given at the listed time points and food intake from a buffet will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Janet C King, PhD, Principal Investigator — Children's Hospital & Research Institute Oakland
Locations (1):
- Children's Hospital Oakland Research Institute, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No